CLINICAL TRIAL: NCT05168293
Title: Comparative Study of the Effect of Entecavir Versus Tenofovir on the Presence of HBV DNA in the Peripheral Blood Mononuclear Cells in Chronic Hepatitis B Patients
Brief Title: Effect of Entecavir Versus Tenofovir on HBV DNA Level in Peripheral Blood Mononuclear Cells
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MAOmar, Principle investigator, Assiut University
Other Study IDs: CSEEVTPHDPBMCCHBP
Record Dates: First submitted 2021-12-13; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Detection of HBV-DNA level in Peripheral Blood Mononuclear cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Entecavir group
  Interventions: Other: Detection of HBV-DNA in Peripheral Blood Mononuclear cells
- Tenofovir group
  Interventions: Other: Detection of HBV-DNA in Peripheral Blood Mononuclear cells

INTERVENTIONS:
Other: Detection of HBV-DNA in Peripheral Blood Mononuclear cells — Detection of HBV-DNA level in Peripheral Blood mononuclear cells

SUMMARY:
Liver disease associated with persistent hepatitis B virus (HBV) infection remains an important public health problem with significant morbidity and mortality. In spite of the existence of an effective vaccine, worldwide approximately 260 million people are chronic HBV surface antigen (HBsAg) carriers and current treatment with interferon and/or nucleoside analogues (NA) is not able to achieve a complete cure.

The key obstacle to HBV eradication is the persistence of HBV DNA in the nuclei of infected hepatocytes, either integrated into the host genome or as a covalently closed circular DNA (cccDNA) episomal form.

While HBV integration is rare and its clinical implications still require investigation, cccDNA plays an essential role in the long-term persistence of HBV infection and can often be detected even following NA therapy and HBsAg seroconversion.

Since quantification of cccDNA in infected hepatocytes requires invasive liver biopsy, more accessible tissues, such as serum or peripheral blood mononuclear cells (PBMCs) have been investigated in different patient populations.

DETAILED DESCRIPTION:
Some reports have shown that cccDNA in serum is a marker of off-treatment virological relapse, whereas others have not found cccDNA in the serum of chronic hepatitis B patients.

Some investigators speculate that PBMCs support HBV replication only partially, with linear and circular relaxed HBV DNA but not cccDNA formed in these cells, while others have detected cccDNA in PBMCs and/or plasma in a variable proportion of patients with chronic and occult HBV infection.

Although hepatocytes are recognized as the main target of HBV infection, HBV and other members of the hepadnaviral family, such as woodchuck hepatitis virus (WHV), have significant lymphotropic properties.

Hepadnaviral infection of lymphoid cells is an important mechanism by whitch virus escapes immune recognition and lymphoid reservoirs, particularly those harbouring drug-resistant HBV, may be the key to develop antiviral resistance.

Positive detection rate of HBV-DNA in neutrophils of chronic hepatitis B patients was 30.95%, After treatment of adefovir, the positive rate of HBV-DNA in neutrophils of chronic hepatitis B patients was 9.52% acting as asource of extrahepatic occult infection.

In liver transplant recipients, HBV in peripheral blood mononuclear cells has been implicated in graft reinfection with a specific lymphoid cell derived viral variant.

Additionally HBV intrauterine infection was primarily caused by maternal to fetal peripheral blood mononuclear cells transport in the second trimester of pregnancy.

The goal of treatment for chronic hepatitis B is to prevent liver disease progression and improve survival by long-term suppression of hepatitis B virus replication in a sustained manner.

A functional HBV cure, defined as a sustained hepatitis B surface antigen loss or seroconversion based on assays with a lower limit of HBsAg detection of 0.05 IU/mL, is a rare event in the natural history of chronic hepatitis B that is associated with a reduced risk of HCC.

Complete HBV cure is defined as an elimination of cccDNA together with durable HBsAg loss and undetectable serum HBV-DNA. Although liver biopsy is needed to measure intrahepatic cccDNA activity, serum biomarkers that reflect cccDNA levels are needed instead. Such as HBV RNA, hepatitis B core-related antigen, and/or quantitative HBsAg have been investigated. Quantification and ratio of large and middle proteins of HBsAg also showed specific patterns across different phases of hepatitis B that would predict the viral activity.

Entecavir (ETV) or tenofovir disoproxititis fumarate (TDF) are recommended as first line therapy in the treatment of naïve chronic hepatitis B because of their higher antiviral potency and higher genetic barriers than other antiviral agents.

In reality, ETV and TDF showed high virological responses of up to 93% and 100%, respectively, and a rare genotypic resistance of only 1.2% and 0%, respectively, during the 5- year follow-up in a cohort study.

In a study evaluating Dynamic changes of HBV-DNA in serum and peripheral blood mononuclear cells of chronic hepatitis B patients, concluded that HBV-DNA exists in PBMCs even after 48 weeks of lamivudine treatment that may reinfect hepatocytes again and cause the relapse of hepatitis.

Coffin., et al 2011; suggested that hepatitis B virus in lymphoid cells may be more resistant to antiviral therapy leading to a differential rate of HBV variant secretion in serum or plasma. Furthermore, HBV quasispecies diversity in liver correlated with antiviral drug resistance and this may have implications for the emergence of dominant resistant HBV variants over time.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic HBV
2. Receiving anti-HB viral therapy (Entecavir or Tenofovir)
3. Compliant on treatment
4. Sustained virological response for at least 2 years

Exclusion Criteria:

1. Patients co-infected with hepatitis C virus
2. Less than 18 years old patients
3. Cirrhotic patients
4. Non compliant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with chronic HBV receiving entecavir or tenofovir with sustained virological response for at least 2 years.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Compare the Effect of Entecavir versus Tenofovir on the Presence of HBV DNA in the Peripheral Blood Mononuclear Cells in Chronic Hepatitis B Patients | 1 week
  Measurment of HBV-DNA level in Peripheral Blood Mononuclear cells

REFERENCES:
- [Result] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Result] Allweiss L, Dandri M. The Role of cccDNA in HBV Maintenance. Viruses. 2017 Jun 21;9(6):156. doi: 10.3390/v9060156. PMID 28635668
- [Result] Tu T, Budzinska MA, Shackel NA, Urban S. HBV DNA Integration: Molecular Mechanisms and Clinical Implications. Viruses. 2017 Apr 10;9(4):75. doi: 10.3390/v9040075. PMID 28394272
- [Result] Lai CL, Wong D, Ip P, Kopaniszen M, Seto WK, Fung J, Huang FY, Lee B, Cullaro G, Chong CK, Wu R, Cheng C, Yuen J, Ngai V, Yuen MF. Reduction of covalently closed circular DNA with long-term nucleos(t)ide analogue treatment in chronic hepatitis B. J Hepatol. 2017 Feb;66(2):275-281. doi: 10.1016/j.jhep.2016.08.022. Epub 2016 Sep 14. PMID 27639844
- [Result] Luo X, Huang Y, Chen Y, Tu Z, Hu J, Tavis JE, Huang A, Hu Y. Association of Hepatitis B Virus Covalently Closed Circular DNA and Human APOBEC3B in Hepatitis B Virus-Related Hepatocellular Carcinoma. PLoS One. 2016 Jun 16;11(6):e0157708. doi: 10.1371/journal.pone.0157708. eCollection 2016. PMID 27310677
- [Result] Singla B, Chakraborti A, Sharma BK, Kapil S, Chawla YK, Arora SK, Das A, Dhiman RK, Duseja A. Levels of hepatitis B virus replicative intermediate in serum samples of chronic hepatitis B patients. Mol Biol Rep. 2014 Jul;41(7):4689-96. doi: 10.1007/s11033-014-3339-7. Epub 2014 Apr 6. PMID 24706057
- [Result] Jun-Bin S, Zhi C, Wei-Qin N, Jun F. A quantitative method to detect HBV cccDNA by chimeric primer and real-time polymerase chain reaction. J Virol Methods. 2003 Sep;112(1-2):45-52. doi: 10.1016/s0166-0934(03)00190-3. PMID 12951212
- [Result] Umeda M, Marusawa H, Seno H, Katsurada A, Nabeshima M, Egawa H, Uemoto S, Inomata Y, Tanaka K, Chiba T. Hepatitis B virus infection in lymphatic tissues in inactive hepatitis B carriers. J Hepatol. 2005 Jun;42(6):806-12. doi: 10.1016/j.jhep.2005.01.016. Epub 2005 Apr 1. PMID 15885350
- [Result] Coffin CS, Osiowy C, Gao S, Nishikawa S, van der Meer F, van Marle G. Hepatitis B virus (HBV) variants fluctuate in paired plasma and peripheral blood mononuclear cells among patient cohorts during different chronic hepatitis B (CHB) disease phases. J Viral Hepat. 2015 Apr;22(4):416-26. doi: 10.1111/jvh.12308. Epub 2014 Sep 9. PMID 25203736
- [Result] Michalak TI. Occult persistence and lymphotropism of hepadnaviral infection: insights from the woodchuck viral hepatitis model. Immunol Rev. 2000 Apr;174:98-111. doi: 10.1034/j.1600-0528.2002.017406.x. PMID 10807510
- [Result] Michalak TI, Mulrooney PM, Coffin CS. Low doses of hepadnavirus induce infection of the lymphatic system that does not engage the liver. J Virol. 2004 Feb;78(4):1730-8. doi: 10.1128/jvi.78.4.1730-1738.2004. PMID 14747538
- [Result] Han Z, Wang J. [Detection and analysis of HBV in polymorphonuclear neutrophils of patients with hepatitis B]. Xi Bao Yu Fen Zi Mian Yi Xue Za Zhi. 2014 Mar;30(3):299-301, 305. Chinese. PMID 24606751
- [Result] Roche B, Feray C, Gigou M, Roque-Afonso AM, Arulnaden JL, Delvart V, Dussaix E, Guettier C, Bismuth H, Samuel D. HBV DNA persistence 10 years after liver transplantation despite successful anti-HBS passive immunoprophylaxis. Hepatology. 2003 Jul;38(1):86-95. doi: 10.1053/jhep.2003.50294. PMID 12829990
- [Result] Shao Q, Zhao X, Yao Li MD. Role of peripheral blood mononuclear cell transportation from mother to baby in HBV intrauterine infection. Arch Gynecol Obstet. 2013 Dec;288(6):1257-61. doi: 10.1007/s00404-013-2893-x. Epub 2013 May 26. PMID 23708388
- [Result] Liaw YF, Kao JH, Piratvisuth T, Chan HL, Chien RN, Liu CJ, Gane E, Locarnini S, Lim SG, Han KH, Amarapurkar D, Cooksley G, Jafri W, Mohamed R, Hou JL, Chuang WL, Lesmana LA, Sollano JD, Suh DJ, Omata M. Asian-Pacific consensus statement on the management of chronic hepatitis B: a 2012 update. Hepatol Int. 2012 Jun;6(3):531-61. doi: 10.1007/s12072-012-9365-4. Epub 2012 May 17. PMID 26201469
- [Result] Tout I, Loureiro D, Mansouri A, Soumelis V, Boyer N, Asselah T. Hepatitis B surface antigen seroclearance: Immune mechanisms, clinical impact, importance for drug development. J Hepatol. 2020 Aug;73(2):409-422. doi: 10.1016/j.jhep.2020.04.013. Epub 2020 Apr 22. PMID 32333923
- [Result] Asselah T, Loureiro D, Boyer N, Mansouri A. Targets and future direct-acting antiviral approaches to achieve hepatitis B virus cure. Lancet Gastroenterol Hepatol. 2019 Nov;4(11):883-892. doi: 10.1016/S2468-1253(19)30190-6. PMID 31609242
- [Result] Pfefferkorn M, Bohm S, Schott T, Deichsel D, Bremer CM, Schroder K, Gerlich WH, Glebe D, Berg T, van Bommel F. Quantification of large and middle proteins of hepatitis B virus surface antigen (HBsAg) as a novel tool for the identification of inactive HBV carriers. Gut. 2018 Nov;67(11):2045-2053. doi: 10.1136/gutjnl-2017-313811. Epub 2017 Sep 26. PMID 28951526
- [Result] You CR, Lee SW, Jang JW, Yoon SK. Update on hepatitis B virus infection. World J Gastroenterol. 2014 Oct 7;20(37):13293-305. doi: 10.3748/wjg.v20.i37.13293. PMID 25309066
- [Result] Liu Y, Corsa AC, Buti M, Cathcart AL, Flaherty JF, Miller MD, Kitrinos KM, Marcellin P, Gane EJ. No detectable resistance to tenofovir disoproxil fumarate in HBeAg+ and HBeAg- patients with chronic hepatitis B after 8 years of treatment. J Viral Hepat. 2017 Jan;24(1):68-74. doi: 10.1111/jvh.12613. Epub 2016 Sep 23. PMID 27658343
- [Result] Ke CZ, Chen Y, Gong ZJ, Meng ZJ, Liu L, Ren ZJ, Zhou ZH. Dynamic changes of HBV DNA in serum and peripheral blood mononuclear cells of chronic hepatitis patients after lamivudine treatment. World J Gastroenterol. 2006 Jul 7;12(25):4061-3. doi: 10.3748/wjg.v12.i25.4061. PMID 16810760
- [Result] Coffin CS, Mulrooney-Cousins PM, Peters MG, van Marle G, Roberts JP, Michalak TI, Terrault NA. Molecular characterization of intrahepatic and extrahepatic hepatitis B virus (HBV) reservoirs in patients on suppressive antiviral therapy. J Viral Hepat. 2011 Jun;18(6):415-23. doi: 10.1111/j.1365-2893.2010.01321.x. PMID 20626626